CLINICAL TRIAL: NCT06209619
Title: Early, Risk Adapted CC-99282 + Rituximab Post CAR T-Cell Therapy for Non-Hodgkin's Lymphoma
Brief Title: CC-99282 + Rituximab Early Post CART for Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nathan Denlinger (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Nathan Denlinger, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23214; NCI-2023-10172 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: B-Cell Non-Hodgkin Lymphoma-Recurrent; Diffuse Large B-Cell Lymphoma-Recurrent; Follicular Lymphoma-Recurrent; High Grade B-Cell Lymphoma-Recurrent; Primary Mediastinal Large B-Cell Lymphoma-Recurrent; Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma-Recurrent; B-Cell Non-Hodgkin Lymphoma-Refractory; Diffuse Large B-Cell Lymphoma-Refractory; Follicular Lymphoma-Refractory; High Grade B-Cell Lymphoma-Refractory; Primary Mediastinal Large B-Cell Lymphoma-Refractory; Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma-Refractory
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rituximab, CC-99282) (Experimental): Patients receive rituximab intravenously (IV) on day 1 of each cycle and CC-99282 orally (PO) once daily (QD) on days 1-14 of each cycle. Treatment repeats every 28 days for up to 6 cycles of rituximab and up to 26 cycles of CC-99282 in the absence of disease progression or unacceptable toxicity. Patients also undergo positron emission tomography (PET)/computed tomography (CT) and collection of blood samples throughout the trial. Patients may undergo biopsy at screening.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Golcadomide; Procedure: Positron Emission Tomography; Biological: Rituximab

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Golcadomide — Given PO
  Other Names: BMS 986369; BMS-986369; BMS986369; CC -99282; CC 99282; CC99282; CelMod CC-99282; Cereblon E3 Ubiquitin Ligase Modulating Agent CC-99282; Cereblon E3 Ubiquitin Ligase Modulating Drug CC-99282; Cereblon Modulator CC-99282
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima

SUMMARY:
This phase I trial tests the safety, side effects and best dose of CC-99282 with rituximab for the treatment of patients who have received chimeric antigen receptor (CAR) T cell therapy for non-Hodgkins lymphoma and in whom have had a sub-optimal response early on to CAR T-cell therapy. Immunotherapy with CC-99282 may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving CC-99282 with rituximab may be a safe and effective treatment option for patients who have received CAR-T cell therapy for relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety profile and maximum tolerated dose (MTD) of early, risk adapted golcadomide (CC-99282)/rituximab for patients with relapsed/refractory (R/R) non-Hodgkin lymphoma (NHL) post-commercial CD19.CAR-T infusion.

SECONDARY OBJECTIVES:

I. To perform a preliminary efficacy analysis of CC-99282 and rituxan early post CD19.CAR-T defined as the progression free survival (PFS) rate at day+150 post initiation of CC-99282.

II. To describe disease response rates in patients with active disease who are treated with CC-99282 + rituximab.

III. To estimate PFS in subjects treated with CC-99282 + rituximab. IV. To estimate the overall survival (OS) in subjects treated with CC-99282 + rituximab.

EXPLORATORY OBJECTIVES:

I. To describe CD19.CAR-T cell expansion and persistence following treatment with CC-99282/rituximab.

II. To evaluate CC-99282/rituximab's effect on CAR T-cells and other immune cell subsets composition and how this effects clinical outcomes.

III. To evaluate CC-99282/rituximab's effect on CAR T-cell and other immune cell subset function and how this effects clinical outcomes.

IV. To evaluate CC-99282/rituximab's effect on the tumor microenvironment (TME) and how this effects clinical outcomes.

OUTLINE: This is a dose-escalation study of CC-99282 in combination with fixed-dose rituximab.

Patients receive rituximab intravenously (IV) on day 1 of each cycle and CC-99282 orally (PO) once daily (QD) on days 1-14 of each cycle. Treatment repeats every 28 days for up to 6 cycles of rituximab and up to 26 cycles of CC-99282 in the absence of disease progression or unacceptable toxicity. Patients also undergo positron emission tomography (PET)/computed tomography (CT) and collection of blood samples throughout the trial. Patients may undergo biopsy at screening.

After completion of study treatment, patients are followed up at days 240, 365, 455, 547, 637, and 730.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information
* Age ≥ 18 years at the time of consent
* Diagnosis of B-cell Non-Hodgkin's lymphoma including either large B-cell lymphoma or follicular lymphoma. Large B-cell subtypes include but are not limited to diffuse large B-cell lymphoma, high grade B-cell lymphoma (except Burkitt's Lymphoma), primary mediastinal B-cell lymphoma, and diffuse large B cell lymphoma transformed from indolent lymphomas
* Eastern Cooperative Oncology Group (ECOG) Score = 0-2
* Prior receipt of standard of care CD19 directed CAR-T cell therapy including axicabtagene ciloleucel, tisagenlecleucel, or lisocabtagene maraleucel
* Pre-CART imaging with PET within 60 days of infusion of CD19.CAR-T. If patient's receive bridging therapy, PET evaluation post bridging therapy is encouraged as part of institutional guidelines, but not mandated for inclusion
* Evidence of objective response on PET/CT at 30 days post CD19.CAR-T infusion (+15/-5 days) compared to baseline pre-CART PET imaging. Objective response in this trial is defined by reduced fludeoxyglucose F-18 (FDG) uptake or reduction in mass size and includes mixed response
* Evidence of sub-optimal response to CD19.CAR-T as defined in this trial by Deauville Score ≥ 3 on PET/CT at 30 days post CART infusion (+15/-5 days)
* Absolute neutrophil count ≥ 7.5 x 10^8/L (obtained within 14 days prior to initiating study treatment)
* Evidence of partial response, though sub-optimal response as determined by persistent MRD positivity. (Example: Deauville Score 1 or 2 is eligible if MRD is positive via clonoseq).

  * Hematological lab values should be without the use of growth factors or transfusion support
  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Hemoglobin ≥ 8 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Hematological lab values should be without the use of growth factors or transfusion support
  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Platelets ≥ 50 x 10^9/L (obtained within 14 days prior to initiating study treatment)

  * Hematological lab values should be without the use of growth factors or transfusion support
  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Estimated glomerular filtration rate (eGFR) (based on chronic kidney disease-epidemiology collaboration [CKD-EPI] * patient's body surface area [BSA] [Du Bois method]/1.73m^2) ≥ 45 ml/min (obtained within 14 days prior to initiating study treatment)

  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Creatinine clearance >60 mL/min (As measured by Crockcroft-Gault equation or direct 24-hour urine measurement)
* Bilirubin ≤ 1.5 × upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level > 2.0 mg/dL if their conjugated bilirubin is < 2.0 × ULN) (obtained within 14 days prior to initiating study treatment)

  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Aspartate aminotransferase (AST) ≤ 3.0 × ULN (obtained within 14 days prior to initiating study treatment)

  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Alanine aminotransferase (ALT) ≤ 3.0 × ULN (obtained within 14 days prior to initiating study treatment)

  * Note: Changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy
* Patients must be able to provide adequate tissue samples for minimal residual disease (MRD) analysis for identification (ID) of baseline tumor deoxyribonucleic acid (DNA). 2 forms of tissue will be acceptable: optional baseline biopsy tissue post CART and prior to initiation of CC-99282, or archival tumor tissue (ex. formalin-fixed paraffin embedded [FFPE] tumor blocks) from a biopsy containing lymphoma prior to CD19.CART
* Fridericia's formula-corrected QT interval (QTcF) < 470 ms
* Patients must be able to swallow/absorb capsules
* Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to enrollment. Pregnancy tests must be medically supervised with a minimum sensitivity of 25mIU/ml. NOTE: a female of childbearing potential is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months, i.e. has had menses at any time in the preceding 24 consecutive months. Documentation of postmenopausal status must be provided. Further information on pregnancy testing and the definition of a female of childbearing potential located in the CC-99282 pregnancy prevention plan document
* Females of childbearing potential are required to use 2 forms of effective methods of contraception or to agree to practice complete abstinence from the time of informed consent, without interruption, at least 28 days before starting CC-99282, throughout the entire duration of CC-99282, during dose interruptions and for at least 6 months and 2 weeks after the last dose of golcadomide (BMS-986369)/CC-99282. The two contraception methods can be comprised one highly effective method and one additional effective (barrier) method. Further information on acceptable methods is located in the CC-99282 pregnancy prevention plan document
* Male subjects with female partners must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of child bearing potential while taking CC-99282, during dose interruptions and for at least 3 months and 2 weeks following the last dose of CC-99282, even if he has undergone a successful vasectomy. Additional information regarding prevention of pregnancy as it pertains to male subjects is contained within the CC-99282 pregnancy prevention plan document
* Subjects with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the experimental regimen are eligible for the trial
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee

Exclusion Criteria:

* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study and lactating females must agree to not breastfeed while taking study drugs)
* Uncontrolled concomitant illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, myocardial infarction within 1 month prior to enrollment, uncontrolled cardiac arrhythmias, uncontrolled seizures, or severe non compensated hypertension (Systolic blood pressure >= 180mmHg or diastolic blood pressure >= 120mmHg)
* Receipt of CD19.CAR-T for any indication other than that stated within the inclusions criteria
* Concomitant use of strong CYP3A inhibitors and inducers. Examples include (but are not limited to):

  * CYP3A inhibitors: atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, and telithromycin.
  * CYP3A inducers: carbamazepine, phenytoin, and rifampin. Patients that are able to come off moderate CYP3A inhibitors/inducers will require a washout period of at least 14 days or 5 half-lives, whichever is shorter, prior to the initiation of study treatment
* Patients who are actively receiving or have received other investigational agents, including herbal supplements, within 2 weeks or 5 half-lives of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | At 30 days post completion of enrollment
  Will describe frequency and nature of adverse events associated with CC-99282 + rituximab post CD19 chimeric antigen receptor (CAR) -T cell therapy using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Maximum tolerated dose | At 30 days post completion of enrollment
  Will use Bayesian Optimal Interval design to define the maximum tolerated dose.

SECONDARY OUTCOMES:
Freedom from progression | At 150 days
  Will utilize baseline positron emission tomography/computed tomography at 30 days post infusion of CD19.CART compared to day+150 PET post initiation of CC-99282.
Number of patients with response to treatment as assessed by PET imaging | At 60 days and 150 days post initiation of CC-99282 and then every 3 months, assessed up to 2 years
  Patients with response to treatment assessed by PET imaging and as defined by the Lugano criteria. Lugano classification is a five-point scale for reporting FDG PET.
Number of patients with response to treatment as assessed by CT imaging | At 60 days and 150 days post initiation of CC-99282 and then every 3 months, assessed up to 2 years
  Patients with response to treatment assessed by CT imaging and as defined by the Lugano criteria. Lugano classification is a five-point scale for reporting FDG PET.
Objective response rate | At 60 days and 150 days post initiation of CC-99282
  Will be calculated with 95% confidence interval.
Progression free survival | Time from initiation of CC-99282 to clinical progression or death, assessed at 150 days and 2 years post infusion of CD19.CAR-T cell therapy
  Will be estimated using the Kaplan-Meier method.
Overall survival | Time from CD19.CAR-T infusion to date of death as a result of any cause, assessed at 150 days and 2 years post infusion of CD19.CAR-T cell therapy
  Will be estimated using the Kaplan-Meier method.
Incidence of adverse events | Up to 2 years
  The frequency and nature of adverse events associated with CC-99282 + rituximab post CD19.CAR-T cell therapy will be described using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Denlinger, DO, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu